CLINICAL TRIAL: NCT06730789
Title: Prospective Comparison of Conservative Treatment Methods in Patients With Lateral Epicondylitis
Brief Title: Conservative Treatment in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yücel Bilgin, MD, Orthopedics and Traumatolody Specialist, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEAH-YB-2020-01
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Athletic Tape

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lateral Epicondylitis (treatment with epicondylitis bandage) (Experimental): Patients with diagnosis of lateral epicondylitis.
  Interventions: Device: Epicondylitis bandage
- Lateral Epicondylitis (treatment with wrist dorsiflexion orthesis) (Experimental): Patients with diagnosis of lateral epicondylitis.
  Interventions: Device: Wrist dorsiflexion splint
- Lateral Epicondylitis (treatment with kinesio tape) (Experimental): Patients with diagnosis of lateral epicondylitis.
  Interventions: Device: Kinesio tape

INTERVENTIONS:
Device: Epicondylitis bandage — A conservative treatment method of lateral epicondylitis.
  Arms: Lateral Epicondylitis (treatment with epicondylitis bandage)
Device: Wrist dorsiflexion splint — A conservative treatment method of lateral epicondylitis.
  Arms: Lateral Epicondylitis (treatment with wrist dorsiflexion orthesis)
Device: Kinesio tape — A conservative treatment method of lateral epicondylitis
  Arms: Lateral Epicondylitis (treatment with kinesio tape)

SUMMARY:
Conservative treatments follow the vast majority of treatments in lateral epicondylitis. In this research, we aimed to elucidate the treatment outcomes of patients via epicondylitis bandage, wrist dorsiflexion splint, and kinesio tape groups by sequential randomization and to compare treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were ≥18 years of age, and had no history of elbow surgery.
* Participants should have pain and sensitivity, with symptom duration less than 12 weeks.
* Patients with a positive result in one of the provocation tests (Maudsley's Test-resisted middle finger extension extensor carpi radialis test), resisted wrist extension, or passive stretching of the wrist extensors (Mill's Test) were included.

Exclusion Criteria:

* Patients under 18 years of age,
* patients who did not consent to participate in the study,
* those who had previous surgery on the elbow,
* presence of cervical spondylosis and radiculopathy,
* presence of endocrine disease,
* presence of autoimmune disease,
* presence of concomitant entrapment neuropathy or polyneuropathy,
* pregnancy,
* presence of systemic inflammatory disease,
* presence of acute trauma,
* presence of deformity in the upper extremity,
* presence of metabolic disease,
* presence of elbow arthritis,
* presence of allergy to kinesio tape and orthoses,
* having received treatment for lateral epicondylitis in the past (exercise, injection, NSAIDs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Visual analog score | Baseline
  Minimum value: 0 Maximum value: 10 Minimum is better.
Visual analog score | At sixth weeks.
  Minimum value: 0 Maximum value:10 Minimum is better.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder Score | Baseline
  Minimum value:0 Maximum value:100 Minimum is better
Disabilities of the Arm, Shoulder Score | At sixth weeks.
  Minimum value:0 Maximum value:100 Minimum is better

OTHER OUTCOMES:
Patient-Rated Tennis Elbow Evaluation Score | Baseline
  Minimum value:0 Maximum value:10 Minimum is better.
Patient-Rated Tennis Elbow Evaluation Score | At sixth weeks.
  Minimum value:0 Maximum value:10 Minimum is better.
hand grip strength | Baseline
  Minimum value: 0 Maximum value: 100 Maximum is better.
hand grip strength | At sixth weeks.
  Minimum value: 0 Maximum value: 100 Maximum is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)